CLINICAL TRIAL: NCT03289624
Title: Support, Health, Activities, Resources, and Education for Persons With Chronic Conditions and Their Family Caregivers: SHARE-Chronic Conditions (SHARE-CC)
Brief Title: SHARE for Persons With Chronic Conditions and Their Family Caregivers
Acronym: SHARE-CC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lost Funding
Sponsor: Benjamin Rose Institute on Aging (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-003
Record Dates: First submitted 2017-08-18; First posted 2017-09-21 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Chronic Health Conditions; Family Caregivers
Keywords: Care Planning; Care Values and Preferences

STUDY DESIGN:
Intervention Model Description: Persons with chronic conditions and their family caregivers will be randomly assigned to a treatment or control group
Who Masked: Participant
Masking Description: No other parties will be masked in the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHARE for Chronic Conditions (Experimental): Six weekly "SHARE for Chronic Conditions (SHARE-CC)" sessions will be conducted in the dyad's home or another location preferred by the participants. A care plan (the SHARE plan) is created that reflects the mutual decisions made by the dyad as a result of their participation in the SHARE-CC program. The SHARE plan is intended to help the caregiver (CG) ensure the PWCC's values and preferences are supported when decisions have to be made in an emergency or in the end stages of the disease. SHARE plans will be documented in a notebook that also contains information on key topics and provides links to local and online resources and services.
  Interventions: Behavioral: SHARE-CC
- Health Coaching (No Intervention): Six 30-minute weekly telephone calls to provide information and education related to the PWCC's conditions and information about services and care options will be conducted.

INTERVENTIONS:
Behavioral: SHARE-CC — Each of the 6 SHARE-CC sessions are structured similarly, starting with the dyad reviewing goals of the session, the CG & PWCC meeting jointly or separately with the SHARE-CC Counselor around session-specific material, & ending with a review of material, addressing questions, & previewing the next session. Sessions titles are: Communication & Health Education; Care Values; Care Preferences; Family, Friends, & Community Resources; Taking care of yourself-taking care of each other; & Take Action Now.
  The SHARE plan will be developed throughout the sessions and reflects the consensus achieved because of participating in SHARE-CC. It is intended to ensure that the PWCC's values & preferences are supported when decisions have to be in the future.
  Arms: SHARE for Chronic Conditions

SUMMARY:
SHARE-CC is an intervention for families facing the challenges of chronic conditions. SHARE-CC (Support, Help, Activities, Resources, and Education) addresses the need for both members of a care dyad to be actively involved in current and future care planning. This intervention aims to increase knowledge of services, improve communication skills and well-being, and facilitate the understanding of care values and preferences in order to create a mutually agreed upon care plan. This intervention will be tested in a randomized control trial.

DETAILED DESCRIPTION:
This project offers a unique and timely opportunity to evaluate the feasibility, acceptability, and efficacy of the SHARE-Chronic Conditions psycho-social intervention. The project will adapt the SHARE intervention, for use with dyads facing the challenges of chronic conditions. The six-session SHARE-CC program will be implemented and evaluated using a randomized controlled trial with 240 participants in northern Ohio, the San Diego and San Francisco Bay areas in California, and New Jersey.

The SHARE-CC intervention addresses the need for a structured approach that targets both members of a care dyad and empowers them to be actively involved in current and future care planning. It has great potential to not only improve psychosocial outcomes for families, but to also impact healthcare decision-making and utilization.

Persons with chronic conditions and their caregivers will be interviewed prior to (Time 1) and after participating (approximately 4 months post-Time 1) in the SHARE-CC intervention or PWCC control group.

ELIGIBILITY:
Inclusion Criteria:

PWCC:

* Living in geographic area of organizations delivering service
* Living at home rather than in an institutional setting
* Have a family CG as defined below
* Confirmed diagnosis of at least one chronic illness (e.g., heart disease, diabetes, COPD, arthritis, kidney disease, stroke, HIV-AIDS, etc.)
* Require assistance with two or more activities of daily living (e.g., shopping, managing medications, dressing) or receives help with complex medical care tasks (e.g., wound care, preparing special meals); and
* Short Blessed error score between 0 and 6 demonstrating normal cognitive function.

For CGs to be eligible

• must be the PWCC's spouse/partner, adult child, in-law, grandchild, step-child, or other close family member who has or will have primary responsibility for providing assistance to the PWCC

Exclusion Criteria:

* Out of geographic areas
* a primary diagnosis of a neurocognitive disorder (e.g. Alzheimer's Disease or related dementia)
* a mental health condition (e.g., schizophrenia, bipolar disorder, major depression)
* a traumatic brain injury,
* intellectual or developmental disability
* individuals experiencing extreme difficulty adjusting and coping to the diagnosis
* individuals in the terminal phase of a chronic condition (i.e., eligible for Hospice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Service Availability Measure (SAM) at 4 months | Measured at baseline and 4 months later
  Asks caregiver if they or their care partner have used any of the 14 services listed (i.e., counseling, support group, respite). If a caregiver has not used a service then their knowledge of the availability of that service is measured
Change from Baseline Emotional-Intimacy Disruptive Behavior Scale at 4 months | Measured at baseline and 4 months later
  Assesses the extent to which a person engaged in eight behaviors during the past month related to withholding or distorting information about their symptoms and feelings to protect their partner from worrying (i.e., how often have you acted more cheerful than you feel?).
Change from Baseline Positive Affect and Negative Affect scales (DQoL) at 4 months | Measured at baseline and 4 months later
  To measures affect, we will use the Positive Affect (6 items) and Negative Affect (9 items) scales of the Dementia Quality of Life Instrument (DQoL; Brod et al., 1999), modified to include only the positive and negative affect subscales in order to reduce response burden

SECONDARY OUTCOMES:
Change from Baseline Dyadic Relationship Scale at 4 months | Measured at baseline and 4 months later
  The Dyadic Relationship Scale includes the Positive Dyadic Interactions and Negative Dyadic Strain subscales.
Change from Baseline Center for Epidemiological Studies Depression Scale (CES-D) at 4 months | Measured at baseline and 4 months later
  A 20-item measure that asks the respondent to rate how often they experienced symptoms of depression in the past week (i.e., restless sleep). Scores range from 0-60, with scores of 16 or more indicating risk for clinical depression
Change from Baseline Health Care Utilization at 4 months | Measured at baseline and 4 months later
  Four single items that measure self-reported physician visits, hospital emergency room visits, and overnight hospital stays in the past four months.
Change from Baseline Disagreements Scale at 4 months | Measured at baseline and 4 months later
  The Disagreements Scale asks respondents five questions about whether they agree or disagree with their care partner about planning, finances, deciding where to go, planning for care, etc.

OTHER OUTCOMES:
Change from Baseline Partners in Health Scale at 4 months | Measured at baseline and 4 months later
  An 11-item scale that measures a person's perception of their level of chronic condition(s) self-management using a 9-point rating scale, with responses ranging from 0=very good to 8=very poor.
Change from Baseline Care Values Scale at 4 months | Measured at baseline and 4 months later
  A 25-item scale that measures the patient's and caregiver's perceptions of the patient's thoughts and feelings about what is most important to them should they need care in the future related to six specific care values (response options include: very important, somewhat important, not so important).
Change from Baseline Leisure and Healthy Behaviors Scale at 4 months | Measured at baseline and 4 months later
  The Leisure Scale measures how often the respondent engaged in 14 different activities (i.e., go shopping, play games). Response options range from 1 (not at all) to 3 (often). The 7-item Healthy Behaviors Scale measures how often the respondent engaged in a variety of health related behaviors (i.e., you got an adequate amount of sleep, you ate too much or too little).
Change from Baseline Preferences for Care Tasks Scale at 4 months | Measured at baseline and 4 months later
  Patients and caregiver's perceptions of the patient's preferences for who they would prefer to help them with 19 care tasks (i.e., shopping, bathing) if they needed assistance in the future. The responses options include: caregiver, other family or friends, and paid providers.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Whitlatch, PhD, Principal Investigator — Benjamin Rose Institute on Aging; Silvia Orsulic-Jeras, Study Director — Benjamin Rose Institute on Aging
Locations (4):
- United States (4):
  - Southern Caregiver Resource Center, San Diego, California
  - Family Caregiver Alliance, San Francisco, California
  - Geriatric Care Consultant, Ridgewood, New Jersey
  - Benjamin Rose Institute on Aging, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Whitlatch, C.J., Clark, P.A., & Schur, D. (2000). COPE: Caregiver Options Program and Evaluation. Final report to nine Cleveland foundations. Benjamin Rose Institute, Cleveland.
- [Background] Battersby, M.W., Ask, A., Reece, M.M., Markwick, M.J., & Collins, J.P. (2003). The Partners in Health scale: The development and psychometric properties of a generic assessment scale for chronic condition self- management. Australian Journal of Primary Health, 9(2 & 3), 41-52.
- [Background] Druley JA, Stephens MA, Coyne JC. Emotional and physical intimacy in coping with lupus: women's dilemmas of disclosure and approach. Health Psychol. 1997 Nov;16(6):506-14. doi: 10.1037//0278-6133.16.6.506. PMID 9386995
- [Background] Bass, D. M., Tausig, M. B., & Noelker, L. S. (1988). Elder impairment,social support and caregiver strain: A framework for understanding support's effects. Journal of Applied Social Sciences, 13, 80-117.
- [Background] Sebern MD, Whitlatch CJ. Dyadic relationship scale: a measure of the impact of the provision and receipt of family care. Gerontologist. 2007 Dec;47(6):741-51. doi: 10.1093/geront/47.6.741. PMID 18192628
- [Background] Whitlatch CJ, Feinberg LF, Tucke SS. Measuring the values and preferences for everyday care of persons with cognitive impairment and their family caregivers. Gerontologist. 2005 Jun;45(3):370-80. doi: 10.1093/geront/45.3.370. PMID 15933277
- [Background] Feinberg LF, Whitlatch CJ. Decision-making for persons with cognitive impairment and their family caregivers. Am J Alzheimers Dis Other Demen. 2002 Jul-Aug;17(4):237-44. doi: 10.1177/153331750201700406. PMID 12184513
- [Background] Zarit SH, Stephens MA, Townsend A, Greene R. Stress reduction for family caregivers: effects of adult day care use. J Gerontol B Psychol Sci Soc Sci. 1998 Sep;53(5):S267-77. doi: 10.1093/geronb/53b.5.s267. PMID 9750575
- [Background] Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978 Mar;19(1):2-21. No abstract available. PMID 649936
- [Background] Mullan JT. The bereaved caregiver: a prospective study of changes in well-being. Gerontologist. 1992 Oct;32(5):673-83. doi: 10.1093/geront/32.5.673. PMID 1427280
- [Background] Aneshensel, C.S., Pearlin, L.I., Mullan, J.T., Zarit, S.H., & Whitlatch,C.J. (1995). Profiles in caregiving: The unexpected career. San Diego, CA: Academic Press
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Brod M, Stewart AL, Sands L, Walton P. Conceptualization and measurement of quality of life in dementia: the dementia quality of life instrument (DQoL). Gerontologist. 1999 Feb;39(1):25-35. doi: 10.1093/geront/39.1.25. PMID 10028768
- [Background] Radloff, L.S. (1977). The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 11, 385-401.
- [Background] Radloff, L.S., & Teri, L. (1986). Use of the Center for Epidemiological Studies-Depression Scale with older adults. Clinical Gerontologist, 5, 119-136.
- [Background] Ritter PL, Stewart AL, Kaymaz H, Sobel DS, Block DA, Lorig KR. Self-reports of health care utilization compared to provider records. J Clin Epidemiol. 2001 Feb;54(2):136-41. doi: 10.1016/s0895-4356(00)00261-4. PMID 11166528
- [Background] Lorig, K., Stewart, A., Ritter, P.L., Gonzalez, V., Laurent, D., & Lynch,J. (1996). Outcome Measures for Health Education and other Health Care Interventions. Thousand Oak, CA: Sage Publications, 24-25